CLINICAL TRIAL: NCT02151643
Title: Study to Evaluate the Efficacy and Safety of PT20 in Subjects With Hyperphosphataemia and Dialysis Dependent Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phosphate Therapeutics (Industry)
Collaborators: Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT20-201
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Hyperphosphataemia
Keywords: Dialysis Dependent Chronic Kidney Disease
MeSH Terms: conditions — Hyperphosphatemia | interventions — Iron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1 - PT20 400 mg tid (Experimental): PT20 400 mg tid (1.2 g/day) administered orally.
  Dosing was initiated with the subject's first meal/snack following receipt of study medication at Visit 7 (Day 1). There was to be no change in dose administration level with respect to each cohort in this study
  Interventions: Drug: PT20
- Group 2 - PT20 800 mg tid (Experimental): PT20 800 mg tid (2.4 g/day) administered orally.
  Dosing was initiated with the subject's first meal/snack following receipt of study medication at Visit 7 (Day 1). There was to be no change in dose administration level with respect to each cohort in this study
  Interventions: Drug: PT20
- Group 3 - PT20 1600 mg tid (Experimental): PT20 1600 mg tid (4.8 g/day) administered orally.
  Dosing was initiated with the subject's first meal/snack following receipt of study medication at Visit 7 (Day 1). There was to be no change in dose administration level with respect to each cohort in this study
  Interventions: Drug: PT20
- Group 4 - PT20 3200 mg tid (Experimental): PT20 3200 mg tid (9.6 g/day) administered orally.
  Dosing was initiated with the subject's first meal/snack following receipt of study medication at Visit 7 (Day 1). There was to be no change in dose administration level with respect to each cohort in this study
  Interventions: Drug: PT20
- Group 5 - Placebo tid (Placebo Comparator): Matched Placebo (for PT20) tid administered orally.
  Dosing was initiated with the subject's first meal/snack following receipt of study medication at Visit 7 (Day 1). There was to be no change in dose administration level with respect to each cohort in this study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PT20 — Modified ferric oxide adipate tablets
  Other Names: Iron (III) oxide adipate; ferric oxide adipate; iron (III) oxide hydroxide adipate; M10L78
  Arms: Group 1 - PT20 400 mg tid; Group 2 - PT20 800 mg tid; Group 3 - PT20 1600 mg tid; Group 4 - PT20 3200 mg tid
Drug: Placebo — Placebo tablets matched to each PT20 dose arm
  Other Names: Matched Placebo for PT20
  Arms: Group 5 - Placebo tid

SUMMARY:
The main purpose of this study is to see whether PT20 can help people with a high level of phosphate in their blood (called Hyperphosphatemia) that are being treated with dialysis for kidney disease.

DETAILED DESCRIPTION:
PT20 represents a mechanism to address many of the limitations associated with current phosphate binding agents. The available clinical and non clinical evidence suggests that PT20 binds phosphate and prevents its uptake more efficiently than other phosphate binding drugs and may therefore either reduce the pill burden associated with controlling phosphate levels, or result in lower phosphate levels with the same pill burden.

The this study is the first to investigate the efficacy and safety of PT20 in subjects with dialysis-dependent chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 90 years
* Subject must have a stable dialysis prescription for at least 28 days prior to start of Screening.
* Subject must have the most recent serum phosphate measurement, taken during the 28 days prior to the start of Screening, of ≥ 4.0 mg/dL and ≤ 8 mg/dL.

Exclusion Criteria:

* Subject's most recent historical pre-dialysis serum bicarbonate value within 14 days prior to the start of Screening (Visit 1) is < 18 mg/dL.
* Subject has, in the opinion of the investigator, severe chronic lung disease and/or carbon dioxide retention.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2014-05-07 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Block, MD, Principal Investigator — Denver Nephrologist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Sampson M, Faria N, Powell JJ; PEACH study investigators. Efficacy and safety of PT20, an iron-based phosphate binder, for the treatment of hyperphosphataemia: a randomized, double-blind, placebo-controlled, dose-ranging, Phase IIb study in patients with haemodialysis-dependent chronic kidney disease. Nephrol Dial Transplant. 2021 Jul 23;36(8):1399-1407. doi: 10.1093/ndt/gfaa116. PMID 32651955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male/female subjects with dialysis dependent CKD on prescribed maintenance haemodialysis 3 times/week for 90d before Screening were recruited and randomised to receive PT20 or placebo. Prior to Screening, all subjects were taking at least 1 OPB for a minimum of 28d mean + serum phosphate level ≥ 4.0 mg/dL and ≤ 8.0 mg/dL for the preceding 28 days.
Pre-assignment Details: Subjects underwent stratified randomisation into 1 of the 4 PT20 dose groups or equivalent placebo group based pre-randomisation serum phosphate level (ratio of 8:8:8:13:13) - serum phosphate < 7.5 mg/dL were deemed to have a lower level of serum phosphate; serum phosphate ≥ 7.5 mg/dL were deemed to have a higher level of serum phosphate.
Groups:
- Group 1 - PT20 400 mg Tid: PT20 400 mg tid (1.2 g/day) administered orally
  PT20: Modified ferric oxide adipate
- Group 2 - PT20 800 mg Tid: PT20 800 mg tid (2.4 g/day) administered orally
  PT20: Modified ferric oxide adipate
- Group 3 - PT20 1600 mg Tid: PT20 1600 mg tid (4.8 g/day) administered orally
  PT20: Modified ferric oxide adipate
- Group 4 - PT20 3200 mg Tid: PT20 3200 mg tid (9.6 g/day) administered orally
  PT20: Modified ferric oxide adipate
- Group 5 - Placebo Tid: Matched Placebo (for PT20) tid administered orally
  Placebo: Placebo tablets matched to each active PT20 dosage arm
Period: Overall Study
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Started | 26 | 25 | 25 | 39 | 38
Completed | 20 | 21 | 21 | 32 | 35
Not Completed | 6 | 4 | 4 | 7 | 3
Not completed — Adverse Event | 2 | 0 | 1 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 1
Not completed — Hyperphosphataemia | 1 | 0 | 0 | 0 | 1
Not completed — High Ferritin levels | 3 | 3 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Safety population - consisting of all subjects who received at least one dose of study medication and had at least one subsequent contact with the Investigator.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid | Total
Number analyzed (Participants) | 24 | 23 | 22 | 36 | 36 | 141
Age, Continuous [Mean (Full Range); unit: years] | 60.4 [26 to 86] | 58.0 [30 to 78] | 60.3 [33 to 84] | 55.9 [26 to 77] | 55.0 [23 to 80] | 57.5 [23 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 11 | 16 | 14 | 58
  Male | 16 | 14 | 11 | 20 | 22 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 8 | 14 | 13 | 53
  Not Hispanic or Latino | 15 | 14 | 14 | 22 | 23 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 1 | 1 | 0 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 0 | 0 | 3
  Black or African American | 7 | 8 | 9 | 12 | 16 | 52
  White | 12 | 11 | 13 | 20 | 16 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 23 | 22 | 36 | 36 | 141
Baseline Serum Phosphate Concentrations [Count of Participants; unit: Participants] — Serum phosphate concentrations were used as stratum for randomisation. The pre-randomisation phosphate levels are summarised.
  Participants
    < 7.5 mg/dL | 13 | 15 | 11 | 20 | 20 | 79
    ≥ 7.5 mg/dL | 11 | 8 | 11 | 16 | 16 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Phosphate Concentration From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: The primary efficacy endpoint was the change in serum phosphate concentration from Baseline (Visit 7, Day 1) to Visit 11 (Day 29). All study specific blood samples were collected, processed and analysed using a central laboratory.
Time Frame: Day 1 to Day 29
Population: Intent-to-Treat (ITT) population.
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 20 | 20 | 20 | 32 | 35
mg/dL | -0.4 [-3.1 to 3.5] | -0.59 [-4.9 to 2.6] | -1.29 [-4.6 to 1.5] | -1.363 [-5.2 to 4.6] | -0.165 [-2.5 to 2.4]
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population - statistical analysis of linear model "fit" using an F-test at the 0.05 level. It was determined that 150 subjects randomised at a ratio of 8:8:8:13:13 (low dose to high dose, placebo) would have >90% power to detect either a statistically significant slope for the dose-response relationship, or, if the relationship was not linear, a statistically significant difference between the highest-dose group and the placebo group, using a two-sided 0.05 significance level; Test type: Other — The primary analysis was a linear model which attempted to explain change from Baseline (Visit 7) to Day 29 (Visit 11) in serum phosphate concentration based on log-transformed dose level (assuming that placebo was equally spaced below the lowest dose level), and stratified by pre-randomisation serum phosphate level (< 7.5 mg/dL or ≥ 7.5 mg/dL). Missing assessments were imputed using the subject's last observed phosphate concentration value (Last Observation Carried Forward [LOCF] imputation); p = 0.784, F-test
Statistical Analysis 2: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population sensitivity analysis using baseline observation carried forward (BOCF) to assess statistical analysis of linear model "fit" using an F-test at the 0.05 level; Test type: Other — Sensitivity analysis of ITT primary analysis using baseline observation carried forward (BOCF) for any missing Day 29 (Visit 11) serum phosphate values; p = 0.905, F-test
Statistical Analysis 3: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population sensitivity analysis using multiple imputation (MI) to assess statistical analysis of linear model "fit" using an F-test at the 0.05 level; Test type: Other — Sensitivity analysis of ITT primary analysis using multiple imputation (MI) for any missing Day 29 (Visit 11) serum phosphate values; p = 0.976, F-test
Statistical Analysis 4: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Per protocol (PP) population sensitivity analysis to assess statistical analysis of linear model "fit" using an F-test at the 0.05 level; Test type: Other — Sensitivity analysis of the primary ITT analysis using the Per Protocol (PP) population; p = 0.914, F-test
Statistical Analysis 5: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population - statistical analysis of the linear model log(PT20 dose)-response relationship to examine whether the linear trend of the change in phosphate level as a function of the log-transformed dose was statistically significant; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.001, linear model - log (dose) - response; Slope = -0.329
Statistical Analysis 6: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - Type 3 tests of fixed effects - treatment group; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - Type 3 tests of fixed effects - visit; Test type: Other; p = 0.436, Mixed Models Analysis
Statistical Analysis 8: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - Type 3 tests of fixed effects - treatment group versus Visit interaction; Test type: Other; p = 0.959, Mixed Models Analysis
Statistical Analysis 9: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - Type 3 tests of fixed effects - baseline serum phosphate concentration; Test type: Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 10: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - Type 3 tests of fixed effects - baseline serum phosphate concentration versus Visit interaction; Test type: Other; p = 0.144, Mixed Models Analysis
Statistical Analysis 11: Comparison: Group 1 - PT20 400 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - mixed model repeated measures for change in serum phosphate concentration; Test type: Other; Mean Difference (Final Values) = 0.117, 97.5% CI 1-sided [upper limit 0.761], Standard Error of Mean 0.2847
Statistical Analysis 12: Comparison: Group 2 - PT20 800 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - mixed model repeated measures for change in serum phosphate concentration; Test type: Other; Mean Difference (Final Values) = 0.007, 97.5% CI 1-sided [upper limit 0.659], Standard Error of Mean 0.2881
Statistical Analysis 13: Comparison: Group 3 - PT20 1600 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - mixed model repeated measures for change in serum phosphate concentration; Test type: Other; Mean Difference (Final Values) = -0.705, 97.5% CI 1-sided [upper limit -0.05], Standard Error of Mean 0.2891
Statistical Analysis 14: Comparison: Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; ITT population supportive analysis - mixed model repeated measures for change in serum phosphate concentration; Test type: Other; Mean Difference (Final Values) = -1.195, 97.5% CI 1-sided [upper limit -0.618], Standard Error of Mean 0.2550

2. Secondary Outcome: Change in Haemoglobin Concentration From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: Descriptive statistics were to be used to summarise values and change from Baseline (Visit 7, Day 1) to Day 29 (Visit 11) in haemoglobin concentration. An analysis of covariance (ANCOVA) was to be used to analyse the changes from Baseline (Visit 7, Day 1) to Visit 11 (Day 29), which were to include the fixed, categorical effects of treatment as well as the continuous, fixed covariates of Baseline concentrations for haemoglobin. Only those subjects with available concentrations for both Baseline (Visit 7, Day 1) and Visit 11 (Day 29) were to be included in this analysis.
Time Frame: Day 1 to Day 29
Population: ITT population.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 19 | 19 | 20 | 31 | 29
g/dL | 0.02 (0.953) | -0.25 (1.085) | -0.22 (0.958) | 0.18 (0.913) | -0.13 (0.892)
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in haemoglobin concentration from Baseline by PT20 dose group; Test type: Other; p = 0.497, ANCOVA
Statistical Analysis 2: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in haemoglobin concentration from Baseline by baseline hemoglobin; Test type: Other; p < 0.001, ANCOVA

3. Secondary Outcome: Change in Serum Ferritin Concentration From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: Descriptive statistics were to be used to summarise values and change from Baseline (Visit 7, Day 1) to Day 29 (Visit 11) in serum ferritin concentration. An analysis of covariance (ANCOVA) was to be used to analyse the changes from Baseline (Visit 7, Day 1) to Visit 11 (Day 29), which were to include the fixed, categorical effects of treatment and week (Visit), as well as the continuous, fixed covariates of Baseline concentrations for serum ferritin. Only those subjects with available concentrations for both Baseline (Visit 7, Day 1) and Visit 11 (Day 29) were to be included in this analysis.
Time Frame: Day 1 to Day 29
Population: ITT population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 20 | 20 | 20 | 31 | 34
ng/mL | 50 (206.23) | 48.8 (231.41) | 10.1 (107.05) | 69.9 (172.85) | -67.0 (181.73)
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in serum ferritin concentration from Baseline by PT20 dose group; Test type: Other; p = 0.243, ANCOVA
Statistical Analysis 2: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in serum ferritin concentration from Baseline by Visit; Test type: Other; p = 0.867, ANCOVA
Statistical Analysis 3: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in serum ferritin concentration from Baseline by baseline serum ferritin concentration; Test type: Other; p = 0.186, ANCOVA

4. Secondary Outcome: Change in Transferrin Saturation From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: Descriptive statistics were to be used to summarise values and change from Baseline (Visit 7, Day 1) to Day 29 (Visit 11) in transferrin saturation. An analysis of covariance (ANCOVA) was to be used to analyse the changes from Baseline (Visit 7, Day 1) to Day 29 (Visit 11), which were to include the fixed, categorical effects of treatment and week, as well as the continuous, fixed covariates of Baseline concentrations for transferrin saturation. Only those subjects with available concentrations for both Baseline (Visit 7, Day 1) and Visit 11 (Day 29) were to be included in this analysis.
Time Frame: Day 1 to Day 29
Population: ITT population.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 20 | 20 | 19 | 29 | 33
percent | 2.20 (8.649) | 0.40 (11.856) | 5.84 (15.178) | -4.59 (14.735) | -0.45 (8.754)
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in transferrin saturation from Baseline by PT20 dose group; Test type: Other; p = 0.068, ANCOVA
Statistical Analysis 2: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in transferrin saturation from Baseline by Visit; Test type: Other; p = 0.013, ANCOVA
Statistical Analysis 3: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in transferrin saturation from Baseline by Baseline Transferrin Saturation; Test type: Other; p < 0.001, ANCOVA

5. Secondary Outcome: Change in Calcium x Phosphate Product From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: Descriptive statistics were to be used to summarise values and change from Baseline (Visit 7, Day 1) to Day 29 (Visit 11) in Calcium x Phosphate Product . An analysis of covariance (ANCOVA) was to be used to analyse the changes from Baseline (Visit 7, Day 1) to Day 29 (Visit 11), which were to include the fixed, categorical effects of treatment, as well as the continuous, fixed covariates of Baseline concentrations for Calcium x Phosphate Product. Only those subjects with available concentrations for both Baseline (Visit 7, Day 1) and Visit 11 (Day 29) were to be included in this analysis. In CKD subjects (Stages 3-5), the clinical recommendation (KDOQI) is that serum calcium x phosphate product should be maintained at < 55 mg^2/dL^2 (4.4 mmol^2 /L^2).
Time Frame: Day 1 to Day 29
Population: ITT population.
Measure: Mean (Standard Deviation); unit: mg^2/dL^2
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 17 | 16 | 16 | 26 | 27
mg^2/dL^2 | -5.515 (13.7966) | -4.035 (13.5196) | -11.127 (15.1683) | -10.996 (19.3057) | -0.778 (10.286)
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in Calcium x Phosphate Product from Baseline by PT20 dose group; Test type: Other; p = 0.004, ANCOVA
Statistical Analysis 2: Comparison: Group 1 - PT20 400 mg Tid vs Group 2 - PT20 800 mg Tid vs Group 3 - PT20 1600 mg Tid vs Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Repeated measures ANCOVA for change in transferrin saturation from Baseline by Baseline Calcium x Phosphate Product; Test type: Other; p < 0.001, ANCOVA

6. Secondary Outcome: Change in Gastrointestinal Symptom Rating System (GSRS) Overall Score From Baseline (Visit 7, Day 1) to Visit 11 (Day 29)
Description: The GSRS assesses the impact of treatment-related GI complications. It includes 15 items divided into 5 subscales (diarrhoea, indigestion, abdominal pain, constipation, and reflux), and uses a seven-grade Likert scale to assess symptoms (1 = no discomfort at all, 7 = very severe discomfort). The total score was calculated as the average score of all 15 items. If data were missing from one or more subscales, the mean of the completed items within the subscale was to be used for the subscale score, provided that more than half of the subscale items were complete. If more than half of the items within a subscale were missing, the subscale score and overall score were also to be defined as missing. The change in overall GSRS score from Baseline (Visit 7, Day 1) to Visit 11 (Day 29) was summarised by treatment and a two-sample t-test was to be used to identify differences between the placebo and PT20 dose groups. The higher the score, the more severe the gastrointestinal symptoms.
Time Frame: Day 1 to Day 29
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
Number analyzed (Participants) | 22 | 21 | 19 | 31 | 34
score on a scale | -0.9 (3.75) | 2.8 (5.97) | 0.4 (9.80) | 1.6 (8.48) | 0.1 (5.16)
Statistical Analysis 1: Comparison: Group 1 - PT20 400 mg Tid vs Group 5 - Placebo Tid; Test type: Other; p = 0.292, paired z-test
Statistical Analysis 2: Comparison: Group 2 - PT20 800 mg Tid vs Group 5 - Placebo Tid; Test type: Other; p = 0.047, paired z-test
Statistical Analysis 3: Comparison: Group 3 - PT20 1600 mg Tid vs Group 5 - Placebo Tid; Test type: Other; p = 0.872, paired z-test
Statistical Analysis 4: Comparison: Group 4 - PT20 3200 mg Tid vs Group 5 - Placebo Tid; Test type: Other; p = 0.288, paired z-test

ADVERSE EVENTS:
Time Frame: All AEs that occurred from the point a subject signed the informed consent form until study completion up to 13 weeks later were to be reported on the eCRF. Any SAE that occurred from the point of a subject signing the informed consent form to within 28 days of the last study visit (as self-reported by subject, up to 17 weeks after informed consent) was to be reported by the Investigator within the eCRF or by fax or telephone within 24 h of awareness of the event.
Description: Subjects were expected to volunteer information about AEs they experienced. The Investigator/designee also questioned the subject at each visit about AEs and recorded these as well as all other AEs apparent. AEs/SAEs were monitored until they were resolved or determined to be due to a subject's on-going condition or inter-current illness.
Arm/Group | Group 1 - PT20 400 mg Tid | Group 2 - PT20 800 mg Tid | Group 3 - PT20 1600 mg Tid | Group 4 - PT20 3200 mg Tid | Group 5 - Placebo Tid
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/22 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/23 | 1/22 | 5/36 | 5/36
Other Adverse Events (participants affected / at risk) | 10/24 | 11/23 | 13/22 | 16/36 | 16/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PT20 400 mg Tid (N=24) | Group 2 - PT20 800 mg Tid (N=23) | Group 3 - PT20 1600 mg Tid (N=22) | Group 4 - PT20 3200 mg Tid (N=36) | Group 5 - Placebo Tid (N=36)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PT20 400 mg Tid (N=24) | Group 2 - PT20 800 mg Tid (N=23) | Group 3 - PT20 1600 mg Tid (N=22) | Group 4 - PT20 3200 mg Tid (N=36) | Group 5 - Placebo Tid (N=36)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (4) | 6 (6) | 2 (2)
Faeces discoloured (Gastrointestinal disorders) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes